CLINICAL TRIAL: NCT05671900
Title: The Efficacy of Sequential Intravesical Gemcitabine and Docetaxel Therapy (GEM/DOCE) in High-risk BCG-naive Patients With Non-muscle Invasive Bladder Cancer (NMIBC)
Brief Title: Gemcitabine and Docetaxel Therapy in High-risk BCG-naive Patients With Non-muscle Invasive Bladder Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Mirko Bakula, PhD, Urologist, Clinical Hospital Centre Zagreb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 81505203284
Record Dates: First submitted 2022-12-20; First posted 2023-01-05 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Non-muscle-invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients (Experimental): All patients receive same intervention throughout the trial.
  Interventions: Drug: Gemcitabine 1000 mg, Docetaxel 37.5g

INTERVENTIONS:
Drug: Gemcitabine 1000 mg, Docetaxel 37.5g — 6 weekly instillations of gemcitabine (1 gram of gemcitabine in 50 ml of sterile water) followed immediately by docetaxel (37.5 mg of docetaxel in 50 mL of saline) and subsequent monthly maintenance installations for those with no evidence of disease.
  Other Names: Sequential intravesical chemotherapy GEM/DOCE

SUMMARY:
Bacillus Calmette-Guerin (BCG) is the standard of care for high-risk patients with non-muscle invasive bladder cancer (NMIBC) after transurethral tumor resection. Since 2012, global BCG shortage encouraged the search of alternative treatment for NMIBC treatment. Intravesical gemcitabine and docetaxel chemotherapy (GEM/DOCE) has shown safety and efficacy in 2 retrospective, single institution cohorts. At our institution, GEM/DOCE has been offered as an option for NMIBC in the treatment of high-risk BCG-naive patients per the protocol adapted from University of Iowa, in shortage situation. Our objective is to evaluate the efficacy of GEM/DOCE therapy.

ELIGIBILITY:
Inclusion Criteria:

* BCG-naive patients with high-risk non-muscle invasive bladder cancer

Exclusion Criteria:

* patients in whome cystectomy is planned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Reccurence free survival | 2 years
  Patients with no bladder cancer reccurence during therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mirko Bakula, Principal Investigator — UHC Zagreb
Locations (1):
- University Hospital Centre Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Yes
Protocol, patients' medical information and results will be shared
Supporting Information: Study Protocol, ICF